CLINICAL TRIAL: NCT06579235
Title: Explorative Proteomics to Ease the Diagnosis of Pediatric Neuroborreliosis
Brief Title: Explorative Proteomics in Pediatric Neuroborreliosis
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Joakim Bloch, Principal Investigator, Medical Doctor, Rigshospitalet, Denmark
Other Study IDs: 9365
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Neuroborreliosis; Facial Palsy; Pediatric Infectious Disease
Keywords: Neuroborreliosis; Pediatric Infectious Disease; Proteomics
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collected in EDTA-tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with neuroborreliosis
  Interventions: Diagnostic Test: Proteomics
- Children without neuroborreliosis
  Interventions: Diagnostic Test: Proteomics

INTERVENTIONS:
Diagnostic Test: Proteomics — All samples of cases (with LNB) and controls (without LNB) will undergo proteomic analyses.

SUMMARY:
This study aims to use proteomic analysis to diagnose Lyme Neuroborreliosis (LNB) in children. Pediatric patients with suspected LNB will be enrolled, and their blood samples will be collected for proteomic analyses. Mass spectrometry will be used to compare protein profiles of LNB-positive and LNB-negative patients. The data will be analyzed by bioinformaticians. The expected impact is to establish a non-invasive, reliable method for early LNB diagnosis to improve patient outcomes.

DETAILED DESCRIPTION:
Objective:

The primary objective of this study is to investigate the utility of proteomic analysis in diagnosing lyme neuroborreliosis (LNB) in children. By identifying specific protein markers associated with LNB (proteomics), the investigators aim to enhance early detection and improve patient outcomes.

Methods:

Participant Recruitment:

The investigators will enroll pediatric patients (aged 1 month to 17 years) presenting with suspected LNB.

Informed consent will be obtained from parents or legal guardians.

Sample Collection:

Peripheral blood samples will be collected from each participant in EDTA tubes. Samples will be processed to carry out proteomic analyses.

Proteomic Analysis:

Mass spectrometry will be employed to compare protein profiles between LNB-positive and LNB-negative patients.

Data Analysis and Presentations:

Protein profiles will be analysed by trained bioinformaticians and mainly presented in volcano plots and heat maps.

Outcome Measures:

Unique proteomic profiles of children with LNB.

Expected Impact:

This study aims to establish a non-invasive and reliable method for diagnosing LNB in children. Early identification will facilitate timely treatment and prevent complications associated with LNB.

ELIGIBILITY:
Inclusion Criteria:

* Presenting at a pediatric ward with facial nerve palsy and/or suspicion of lyme neuroborreliosis
* Parental informed consent

Exclusion Criteria:

* Parents or legal guardians unable to understand given information or comply with study criteria
* Patient unable to cooperate to study procedures (blood sample)
* Unclear etiology after lumbar puncture

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children aged 1 month to 17 years presenting at pediatric wards in the capital region of Denmark with facial nerve palsy and/or suspicion of lyme neuroborreliosis.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-12-10 (Estimated)

PRIMARY OUTCOMES:
Protein concentrations | An average of 2 years from enrollment
  A matrix of concentrations of various proteins potentially relevant in diagnosing lyme neuroborreliosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Department of Children and Adolescents, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No